CLINICAL TRIAL: NCT04933162
Title: UC Cohort - The Influence of Diet on Host Physiology and Disease Across Diverse Human Gut Microbiotas
Brief Title: UC Cohort - The Influence of Diet on Gut Microbiotas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Laura E. Raffals, M.D, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20-012389
Record Dates: First submitted 2021-06-15; First posted 2021-06-21 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Diet, Protein-Restricted

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Protein and Low Fiber Group (Experimental): Subjects will consume a high protein and low fiber diet for 8 weeks
  Interventions: Dietary Supplement: High Protein and Low Fiber Diet
- Low Protein and High Fiber Group (Experimental): Subjects will consume a low protein and high fiber diet for 8 weeks
  Interventions: Dietary Supplement: Low Protein and High Fiber Diet

INTERVENTIONS:
Dietary Supplement: High Protein and Low Fiber Diet — Protein intake will be increased to be >40% calories from protein, and the fiber intake will remain <15gm/day.
  Arms: High Protein and Low Fiber Group
Dietary Supplement: Low Protein and High Fiber Diet — Increase fiber intake up to 40gms of fiber with a requirement to increase at least 15gms above baseline fiber, with 50-75% of total fiber intake from psyllium husk. Subjects will be allowed to slowly increase fiber every two days to reach goal by end of week 1. The total protein will be reduced to <10% total calories from protein.
  Arms: Low Protein and High Fiber Group

SUMMARY:
The purpose of this research is to determine if different diets have different effects on the inflammation in the colon.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 years old
2. Ability to give informed consent
3. Diagnosis of ulcerative colitis
4. Moderate UC disease activity defined by a Mayo Score of >6 with endoscopic score of 2
5. On a baseline diet characterized by:

   * Fiber intake of < 15g/day
   * > 18% of daily calories from protein

Exclusion Criteria:

1. Prior history of gastrointestinal surgeries (except appendectomy and cholecystectomy)
2. Use of tobacco products within the past 6 months (since nicotine may affect intestinal permeability)
3. Use of NSAIDs or aspirin and unable or unwilling to stop taking two weeks prior to permeability test and for the duration of the study
4. Use of osmotic laxatives and unable or unwilling to stop taking one week prior to permeability test and for the duration of the study
5. Use of oral corticosteroids and unable or unwilling to stop use of oral corticosteroids within the previous 2 weeks and for the duration of the study
6. Multiple dietary restrictions or unable/unwilling to alter dietary protein or dietary fiber.
7. Unwilling to stop ingestion of alcohol and artificial sweeteners such as Splenda™ (sucralose), Nutrasweet™ (aspartame), sorbitol, xylitol, lactulose, or mannitol 2 days before and during the permeability testing days, e.g. foods to be avoided are sugarless gums or mints and diet beverages
8. Unwilling to stop stenuous exercise (running >5 miles or equivalent) one week prior to the permeability tests
9. Bowel preparation for colonoscopy less than one week prior to completion of the first stool kit and permeability test and flexible sigmoidoscopy and upper endoscopy
10. Pregnancy or plan to become pregnant during the study time frame
11. Vulnerable adult
12. Known bleeding disorders or takes medications that increase risk of bleeding from mucosal biopsies
13. Use of oral antibiotic(s) within the past 4 weeks (can be enrolled after 4-week washout period)
14. Use of commercial probiotic formulations and unwilling to stop for the duration of the study
15. Diagnosis of diabetes
16. Any other disease(s), condition(s) or habits(s) that would interfere with completion of study, or in the judgment of the investigator would potentially interfere with compliance to this study or would adversely affect study outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
Decrease in endoscopic Mayo score for ulcerative colitis inflammation | 8 weeks
  Measured from unprepped, non-sedated flexible sigmoidoscopy by decrease in Mayo score with a decrease of at least 1 point on the endoscopic subscore or absolute endoscopic subscore of 0-1).
Clinical remission derived from patient reported outcomes | 8 weeks
  Defined as a Mayo score ≤2 and no sub-scores with a value greater than 1 is a secondary endpoint. This what the patient reports for stool frequency and reporting of any blood in the stool

SECONDARY OUTCOMES:
Intestinal inflammation determined from blood and stool samples | 8 weeks
  Measures C-reactive protein from blood samples and fecal calprotectin from stool samples
Urinary excretion of lactulose and 13C-Mannitol | 8 weeks
  Small Bowel and Colonic Permeability by Urinary Excretion of Lactulose and 13C-Mannitol after Oral Ingestion of lactulose and 13C mannitol (5:1 ratio by mass). The 0-2h urine most closely reflects small intestinal permeability and 8-24h urine reflects colonic permeability. HPLC-tandem mass spectrometry will be used for detection of the sugars. The results will be expressed as the ratio of percentage excretion of the ingested dose of lactulose and mannitol in urine.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Raffals, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials